CLINICAL TRIAL: NCT04470661
Title: Diagnostic Accuracy of Point-of-Care Ultrasound in the Etiology of Acute Kidney Injury
Brief Title: Point-of-care Ultrasound for Acute Kidney Injury
Status: Completed | Type: Observational
Sponsor: Mehmet Ali Aslaner (Other)
Responsible Party: Sponsor-Investigator, Mehmet Ali Aslaner, Assoc. Prof., Gazi University
Organization: Gazi University (Other)
Other Study IDs: GaziU-2
Record Dates: First submitted 2020-07-09; First posted 2020-07-14 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ultrasonography — Point-of-care ultrasound:
  1. Kidney length and echogenity,
  2. Bladder scanning
  3. VCI measures
  4. Lung B lines and effusion
  5. Cardiac measurements; EF, TAPSE, TR Vmax, Diameters, LV filling pressures

SUMMARY:
It is aimed to determine prerenal, renal and postrenal diagnoses of patients with acute kidney injury with POCUS performed in the emergency department. Patients who presented to the emergency department and who have acute kidney injury (AKI) according to the KDIGO criteria will be evaluated and patients diagnosed with AKI will be included in the study. The diagnostic accuracy of POCUS with the AKI etiologies of the patients will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

• AKI diagnosis according to KDIGO criteria

Exclusion Criteria:

* Patients with end stage renal failure,
* Failure to perform POCUS in the first two hours of presentation of patient,
* Those with renal malignancy,
* Pregnant women,
* Renal transplantation patients,
* Patients with a single kidney,
* Those with polycystic kidney disease,
* Patients with nephrostomy,
* Patients who are referred from another center,
* Unable to perform adequate imaging,
* Patients who do not give consent for the study will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute kidney injury diagnosed in the ED.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
The diagnostic accuracy of POCUS in the patients with AKI | One year

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Aslaner, MD, Principal Investigator — Gazi University
Locations (1):
- Gazi University Facaulty of Medicine, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided